CLINICAL TRIAL: NCT04619342
Title: Safety and Efficacy of GSMs-TACE Combined With Surgical Resection in the Treatment of Hepatocellular Carcinoma (HCC) With Type III Portal Vein Tumor Thrombus (PVTT): A Single Center, Open, Randomized Controlled Trial.
Brief Title: Safety and Efficacy of GSMs-TACE Combined With Surgical Resection in the Treatment of Hepatocellular Carcinoma (HCC) With Type III Portal Vein Tumor Thrombus (PVTT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20304-0-01
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma (HCC) With Type III Portal Vein Tumor Thrombus (PVTT)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSMs-TACE+ Surgical Resection Group (Experimental): After TACE using epirubicin and GSMs (150-350μm or 350-560μm), patients that meet certain criteria will receive surgical resection of PVTT, as specified per protocol.
  Interventions: Device: GSMs-TACE; Procedure: Surgical Resection
- GSMs-TACE Group (Active Comparator): Patients will receive TACE using epirubicin and GSMs (150-350μm or 350-560μm), as specified per protocol.
  Interventions: Device: GSMs-TACE

INTERVENTIONS:
Device: GSMs-TACE — TACE using epirubicin (30-40mg/m2) and gelatin sponge microspheres (150-350μm or 350-560μm)
  Other Names: TACE
Procedure: Surgical Resection — Surgical Resection of PVTT
  Arms: GSMs-TACE+ Surgical Resection Group

SUMMARY:
A Single center, Open, Randomized Controlled Trial Evaluating the Safety and Efficacy of GSMs-TACE Combined with Surgical Resection in the Treatment of Hepatocellular Carcinoma (HCC) with Type III Portal Vein Tumor Thrombus (PVTT).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of HCC with PVTT involving the main portal vein, i.e. Type III PVTT according to Cheng's classification.
2. Confirmed abundant blood supply of tumor thrombus using Computed Tomography (CT) and Magnetic Resonance Imaging (MRI).
3. The tumor must be surgically resectable.
4. ECOG Performance Status 0-2.
5. Adequate liver function (Child-Pugh class A)
6. Life expectancy ≥ 3 months
7. Previous physical ablation is allowed.
8. Age 18 to 75 years
9. Able to sign and provide written informed consent.

Exclusion Criteria:

1. Patients previously took oral molecular targeted drug or received immunotherapy.
2. Patients with arteriovenous fistula.
3. Severe active infection >grade 2 (except for Hepatitis B and C infection).
4. Concomitant malignant tumors in other organs.
5. Presence of severe cardiac, lung or kidney disease.
6. Pregnant or breast-feeding woman.
7. Patients with severe neuropathy and unable to report therapeutic effects.
8. Patients with severe atherosclerosis.
9. Patients with AIDS.
10. Severe hemorrhage of digestive tract within the 4 weeks prior to enrolment.
11. Severe thrombogenesis or embolic event within the 6 months prior to enrolment.
12. Currently enrolled or going to enroll in any other clinical trials.
13. Subject is not suitable to participate in the study as judged by investigator (poor patient compliance, inability to follow up).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | 6 months
  PFS is defined as the time from Day 1 of treatment until the progression of a target lesion or the appearance of new lesions.

SECONDARY OUTCOMES:
Median Overall Survival (mOS) | 2 years
Overall Survival | 3, 6, 12 and 18 months
Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuewei Zhang, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Changgung Hospital, Beijing, China